CLINICAL TRIAL: NCT00180102
Title: AML2003 - Randomized Comparison Between Standard-Therapy and Intensified Therapy for Adult Acute Myeloid Leukemia Patients <= 60 Years. A Prospective, Randomized, Multi-center Therapy-Optimizing-Study.
Brief Title: AML2003 - Standard-Therapy vs Intensified Therapy for Adult Acute Myeloid Leukemia Patients <= 60 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Prof. Dr. G. Ehninger, Medical Department I, University Hospital Dresden
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MK1-95
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Leukemia, Nonlymphocytic, Acute
Keywords: acute myeloid leukemia; risk adapted treatment; early allogeneic stem cell transplantation; autologous stem cell transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute

INTERVENTIONS:
Drug: Cytarabine vs. Cytarabine+Amsacrine+Mitoxantrone
Procedure: early allogeneic PBSCT within induction therapy
Procedure: autologous PBSCT

SUMMARY:
AML2003 is a prospective randomized trial, to investigate the value of early allogeneic stem cell transplantation in aplasia after induction therapy for high risk patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
AML2003 is a prospective randomized trial, to investigate the value of early allogeneic stem cell transplantation in aplasia after induction therapy for high risk patients with acute myeloid leukemia. A rapid analysis of risk-factors (cytogenetics, FLT3 status, clearance of blasts after first induction) and the donor situation is of utmost importance. For this "fast search" diagnostic, which is accomplished in all enclosed patients, significant resources are provided, to take the load off the participating centers. Furthermore, the relevance of autologous transplantation and the benefit of additional substances within the postremission therapy such as m-AMSA or mitoxantrone will be investigated. There is an up-front randomisation in four therapy arms with two cross-classifying factors of two stages (intensified vs. standard therapy and Ara C vs. Ara C+ mitoxantrone + m-AMSA). Thus, the intergroup treatment schedule of the German Competence Network is integrated into the AML2003 study as a central element and 25% of the patients are treated accordingly. In the intensified therapy arms a risk-adapted and priority-based therapy is implemented, including early allogeneic and consolidating autologous stem cell transplantation, respectively. In addition to the clinical questions , a detailed concomitant research program was initiated for the AML2003 study, to get a better view of the heterogeneity of AML and to open new ways for "custom-made" therapies.

ELIGIBILITY:
Inclusion Criteria:

* de novo or secondary acute myeloid leukemia FAB-subtypes M0-M2 and M4-M7
* de novo or secondary myelodysplastic syndrome WHO-type RAEB-2
* age 16 to 60 years
* written informed consent

Exclusion Criteria:

* severe comorbidities
* severe, uncontrolled complications of the leukemia
* prior therapy for AML/MDS
* other simultaneous hematological malignancies
* HIV-Infection
* known allergies against study medication
* pregnancy
* missing written informed consent

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2003-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
overall survival
relapse-free survival

SECONDARY OUTCOMES:
complete remission rate after induction therapy
subgroup-analyses within the primary outcomes according to different risk factors
development of explanatory proportional hazard-models

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Ehninger, MD, Principal Investigator — University Hospital Carl Gustav Carus Dresden
Locations (1):
- Medical Department I, University Hospital Carl Gustav Carus, Dresden, Germany

REFERENCES:
- [Derived] Kunadt D, Stasik S, Metzeler KH, Rollig C, Schliemann C, Greif PA, Spiekermann K, Rothenberg-Thurley M, Krug U, Braess J, Kramer A, Hochhaus A, Scholl S, Hilgendorf I, Brummendorf TH, Jost E, Steffen B, Bug G, Einsele H, Gorlich D, Sauerland C, Schafer-Eckart K, Krause SW, Hanel M, Hanoun M, Kaufmann M, Wormann B, Kramer M, Sockel K, Egger-Heidrich K, Herold T, Ehninger G, Burchert A, Platzbecker U, Berdel WE, Muller-Tidow C, Hiddemann W, Serve H, Stelljes M, Baldus CD, Neubauer A, Schetelig J, Thiede C, Bornhauser M, Middeke JM, Stolzel F; A. M. L. Cooperative Group (AMLCG), Study Alliance Leukemia (SAL). Impact of IDH1 and IDH2 mutational subgroups in AML patients after allogeneic stem cell transplantation. J Hematol Oncol. 2022 Sep 5;15(1):126. doi: 10.1186/s13045-022-01339-8. PMID 36064577
- [Derived] Kunadt D, Kramer M, Dill C, Altmann H, Wagenfuhr L, Mohr B, Thiede C, Rollig C, Schetelig J, Bornhauser M, Schaich M, Stolzel F. Lysyl oxidase expression is associated with inferior outcome and Extramedullary disease of acute myeloid leukemia. Biomark Res. 2020 Jun 12;8:20. doi: 10.1186/s40364-020-00200-9. eCollection 2020. PMID 32537166
- [Derived] Heidrich K, Thiede C, Schafer-Eckart K, Schmitz N, Aulitzky WE, Kramer A, Rosler W, Hanel M, Einsele H, Baldus CD, Trappe RU, Stolzel F, Middeke JM, Rollig C, Taube F, Kramer M, Serve H, Berdel WE, Ehninger G, Bornhauser M, Schetelig J; Study Alliance Leukemia (SAL). Allogeneic hematopoietic cell transplantation in intermediate risk acute myeloid leukemia negative for FLT3-ITD, NPM1- or biallelic CEBPA mutations. Ann Oncol. 2017 Nov 1;28(11):2793-2798. doi: 10.1093/annonc/mdx500. PMID 28945881
- [Derived] Rollig C, Bornhauser M, Kramer M, Thiede C, Ho AD, Kramer A, Schafer-Eckart K, Wandt H, Hanel M, Einsele H, Aulitzky WE, Schmitz N, Berdel WE, Stelljes M, Muller-Tidow C, Krug U, Platzbecker U, Wermke M, Baldus CD, Krause SW, Stolzel F, von Bonin M, Schaich M, Serve H, Schetelig J, Ehninger G. Allogeneic stem-cell transplantation in patients with NPM1-mutated acute myeloid leukemia: results from a prospective donor versus no-donor analysis of patients after upfront HLA typing within the SAL-AML 2003 trial. J Clin Oncol. 2015 Feb 10;33(5):403-10. doi: 10.1200/JCO.2013.54.4973. Epub 2014 Dec 29. PMID 25547501
- [Derived] Herold T, Metzeler KH, Vosberg S, Hartmann L, Rollig C, Stolzel F, Schneider S, Hubmann M, Zellmeier E, Ksienzyk B, Jurinovic V, Pasalic Z, Kakadia PM, Dufour A, Graf A, Krebs S, Blum H, Sauerland MC, Buchner T, Berdel WE, Woermann BJ, Bornhauser M, Ehninger G, Mansmann U, Hiddemann W, Bohlander SK, Spiekermann K, Greif PA. Isolated trisomy 13 defines a homogeneous AML subgroup with high frequency of mutations in spliceosome genes and poor prognosis. Blood. 2014 Aug 21;124(8):1304-11. doi: 10.1182/blood-2013-12-540716. Epub 2014 Jun 12. PMID 24923295
- [Derived] Schaich M, Parmentier S, Kramer M, Illmer T, Stolzel F, Rollig C, Thiede C, Hanel M, Schafer-Eckart K, Aulitzky W, Einsele H, Ho AD, Serve H, Berdel WE, Mayer J, Schmitz N, Krause SW, Neubauer A, Baldus CD, Schetelig J, Bornhauser M, Ehninger G. High-dose cytarabine consolidation with or without additional amsacrine and mitoxantrone in acute myeloid leukemia: results of the prospective randomized AML2003 trial. J Clin Oncol. 2013 Jun 10;31(17):2094-102. doi: 10.1200/JCO.2012.46.4743. Epub 2013 Apr 29. PMID 23630210
- [Derived] Buchner T, Schlenk RF, Schaich M, Dohner K, Krahl R, Krauter J, Heil G, Krug U, Sauerland MC, Heinecke A, Spath D, Kramer M, Scholl S, Berdel WE, Hiddemann W, Hoelzer D, Hehlmann R, Hasford J, Hoffmann VS, Dohner H, Ehninger G, Ganser A, Niederwieser DW, Pfirrmann M. Acute Myeloid Leukemia (AML): different treatment strategies versus a common standard arm--combined prospective analysis by the German AML Intergroup. J Clin Oncol. 2012 Oct 10;30(29):3604-10. doi: 10.1200/JCO.2012.42.2907. Epub 2012 Sep 10. PMID 22965967
- [Derived] Pfirrmann M, Ehninger G, Thiede C, Bornhauser M, Kramer M, Rollig C, Hasford J, Schaich M; Study Alliance Leukaemia (SAL). Prediction of post-remission survival in acute myeloid leukaemia: a post-hoc analysis of the AML96 trial. Lancet Oncol. 2012 Feb;13(2):207-14. doi: 10.1016/S1470-2045(11)70326-6. Epub 2011 Dec 22. PMID 22197676